CLINICAL TRIAL: NCT04033562
Title: The Analgesic Efficacy of Continuous Sub-fascial Bupivacaine Infusion and Lidocaine Patches in Post-cesarean Patients With Opiate Use Disorder: A Comparative Efficacy Analysis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: limited enrollment and unable to enroll subjects to reach statistical significance
Sponsor: WellSpan Health (Other)
Collaborators: Ambu A/S (Industry); York Opioid Collaborative, Pennsylvania (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1351850
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Opioid-use Disorder; Opioid Use; Opioid Dependence; Opioid Abuse; Medication Assisted Treatment; Infusion Catheter, Wound; Lidopatch; Ambu ACTion; Pregnancy Related; Cesarean Section
MeSH Terms: conditions — Opioid-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Lidoderm patch (Active Comparator): Participants will receive a topical 3.6% Lidocaine/1.25% Menthol patch at the time of their Cesarean section. Patches will be replaced every 12 hours for a total of 60 hours.
  Interventions: Drug: Lidocaine patch
- Infusion pump (Active Comparator): Participants will undergo placement of Ambu ACTion drug delivery system at the time of Cesarean delivery. 0.125% of bupivacaine will be infused at a rate of 8cc/hr for a total of 48-60hrs post-operatively.
  Interventions: Device: Ambu ACTion pump, 0.125% bupivacaine at 8cc/hr

INTERVENTIONS:
Drug: Lidocaine patch — Lidocaine patch will be applied at time of Cesarean delivery for post-operative pain control.
  Arms: Lidoderm patch
Device: Ambu ACTion pump, 0.125% bupivacaine at 8cc/hr — Infusion pump will be placed at time of Cesarean delivery for post-operative pain control.
  Arms: Infusion pump

SUMMARY:
Pregnant women with a history of opioid use disorder, chronic opioid use or those who are on medication assisted treatment will be randomly assigned to receive either a sub-fascial continuous infusion of bupivacaine or lidocaine/menthol patch after Cesarean delivery. Post-operative pain scores and opioid usage in the post-operative period will be recorded.

DETAILED DESCRIPTION:
Pregnant women 18 years or older with a history of chronic opioid use, opioid use disorder or women on medication assisted treatment (MAT), will be enrolled in the study and randomly assigned to one of two study groups. The first group will receive a Lidocaine/Menthol patch at the time of her Cesarean delivery, the second will receive placement of the Ambu ACTion infusion pain system at the time of the C-section. This device will be set up to infuse 0.125% of bupivacaine for 48-60hrs postoperatively at a rate of 8cc/hr.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* undergoing a Cesarean delivery via a transverse incision at York Hospital labor and delivery
* Documented history of chronic opioid use or documented OUD, or currently utilizing medically assisted treatment (MAT)

Exclusion Criteria:

* Patients with a history of clinically significant cardiovascular, hepatic, or renal disease
* Non-English speaking
* Allergy to bupivacaine, lidocaine, zinc, silver or menthol
* Unable to consent, due to lack of decisional capacity or need for emergent Cesarean delivery
* History of glucose-6-phosphate deficiency
* Use of anti-arrhythmic drugs such as tocainide or mexiletine

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Pain scores | post-operative until 60 hours postpartum
  Post-operative pain scores using the visual analog scale (a scale that measures pain in 1 unit increments on a scale 0-10 with 0 being "no pain at all" and 10 being "the worst pain imaginable"

SECONDARY OUTCOMES:
Rescue opioid consumption | post-operative until 60 hours postpartum
  Total opioid consumption in MME (morphine milligram equivalent) that patients received post-operatively
Survey of nursing staff | between 48-60 hours post-Cesarean delivery
  1-item questionnaire to assess whether nursing felt that patient benefited from therapy. A Likert scale will be used (strongly agree, agree, neutral, disagree, strongly disagree)
Patient survey | between 48-60 hourrs post-Cesarean delivery
  2-item questionnaire to assess whether patient felt like she benefited from therapy and whether she would elect to use it again in a future C-section. A Likert scale will be used (strongly agree, agree, neutral, disagree, strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Burcher, MD, Principal Investigator — WellSpan Health Ob-Gyn Residency Program Director
Locations (1):
- WellSpan Health York Hospital, York, Pennsylvania, United States

REFERENCES:
- [Background] Ranta PO, Ala-Kokko TI, Kukkonen JE, Ohtonen PP, Raudaskoski TH, Reponen PK, Rawal N. Incisional and epidural analgesia after caesarean delivery: a prospective, placebo-controlled, randomised clinical study. Int J Obstet Anesth. 2006 Jul;15(3):189-94. doi: 10.1016/j.ijoa.2006.02.003. PMID 16798442
- [Background] Fredman B, Shapiro A, Zohar E, Feldman E, Shorer S, Rawal N, Jedeikin R. The analgesic efficacy of patient-controlled ropivacaine instillation after Cesarean delivery. Anesth Analg. 2000 Dec;91(6):1436-40. doi: 10.1097/00000539-200012000-00025. PMID 11093995
- [Background] Givens VA, Lipscomb GH, Meyer NL. A randomized trial of postoperative wound irrigation with local anesthetic for pain after cesarean delivery. Am J Obstet Gynecol. 2002 Jun;186(6):1188-91. doi: 10.1067/mob.2002.122984. PMID 12066096
- [Background] Kainu JP, Sarvela J, Halonen P, Puro H, Toivonen HJ, Halmesmaki E, Korttila KT. Continuous wound infusion with ropivacaine fails to provide adequate analgesia after caesarean section. Int J Obstet Anesth. 2012 Apr;21(2):119-24. doi: 10.1016/j.ijoa.2011.12.009. Epub 2012 Feb 16. PMID 22341892
- [Background] Lalmand M, Wilwerth M, Fils JF, Van der Linden P. Continuous Ropivacaine Subfascial Wound Infusion Compared With Intrathecal Morphine for Postcesarean Analgesia: A Prospective, Randomized Controlled, Double-Blind Study. Anesth Analg. 2017 Sep;125(3):907-912. doi: 10.1213/ANE.0000000000001892. PMID 28368941
- [Background] Jolly C, Jathieres F, Keita H, Jaouen E, Guyot B, Torre A. Cesarean analgesia using levobupivacaine continuous wound infiltration: a randomized trial. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:125-30. doi: 10.1016/j.ejogrb.2015.08.023. Epub 2015 Aug 25. PMID 26366789
- [Background] Guidelines for laparoscopic surgery during pregnancy. Society of American Gastrointestinal Endoscopic Surgeons (SAGES). Surg Endosc. 1998 Feb;12(2):189-90. No abstract available. PMID 9479743
- [Background] Habib AS, Polascik TJ, Weizer AZ, White WD, Moul JW, ElGasim MA, Gan TJ. Lidocaine patch for postoperative analgesia after radical retropubic prostatectomy. Anesth Analg. 2009 Jun;108(6):1950-3. doi: 10.1213/ane.0b013e3181a21185. PMID 19448228
- [Background] Kwon YS, Kim JB, Jung HJ, Koo YJ, Lee IH, Im KT, Woo JS, Im KS. Treatment for postoperative wound pain in gynecologic laparoscopic surgery: topical lidocaine patches. J Laparoendosc Adv Surg Tech A. 2012 Sep;22(7):668-73. doi: 10.1089/lap.2011.0440. Epub 2012 Aug 3. PMID 22861076
- [Background] Khanna M, Peters C, Singh JR. Treating pain with the lidocaine patch 5% after total knee arthroplasty. PM R. 2012 Sep;4(9):642-6. doi: 10.1016/j.pmrj.2012.06.003. Epub 2012 Jul 28. PMID 22841969
- [Background] Bajwa SJ, Kaur J. Clinical profile of levobupivacaine in regional anesthesia: A systematic review. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):530-9. doi: 10.4103/0970-9185.119172. PMID 24249993
- [Background] Brower MC, Johnson ME. Adverse effects of local anesthetic infiltration on wound healing. Reg Anesth Pain Med. 2003 May-Jun;28(3):233-40. doi: 10.1053/rapm.2003.50050. No abstract available. PMID 12772142
- [Background] Tam KW, Chen SY, Huang TW, Lin CC, Su CM, Li CL, Ho YS, Wang WY, Wu CH. Effect of wound infiltration with ropivacaine or bupivacaine analgesia in breast cancer surgery: A meta-analysis of randomized controlled trials. Int J Surg. 2015 Oct;22:79-85. doi: 10.1016/j.ijsu.2015.07.715. Epub 2015 Aug 12. PMID 26277531
- [Background] Scott NB. Wound infiltration for surgery. Anaesthesia. 2010 Apr;65 Suppl 1:67-75. doi: 10.1111/j.1365-2044.2010.06241.x. PMID 20377548
- [Background] Cobb B, Liu R, Valentine E, Onuoha O. Breastfeeding after Anesthesia: A Review for Anesthesia Providers Regarding the Transfer of Medications into Breast Milk. Transl Perioper Pain Med. 2015;1(2):1-7. PMID 26413558
- See also: Bupivacaine hydrochloride — https://www.accessdata.fda.gov/drugsatfda_docs/label/2010/071165s020lbl.pdf
- See also: Wide-ranging online data for epidemiologic research (WONDER) — http://wonder.cdc.gov